CLINICAL TRIAL: NCT06403878
Title: Prospective, Single-arm, Phase II Study of Nab-paclitaxel Plus Carboplatin in Combination With Sintilimab for Neoadjuvant Therapy in Elderly, Locally Advanced, Resectable Esophageal Squamous Cell Carcinoma.
Brief Title: Safety and Efficacy of Neoadjuvant Immunochemotherapy in Elderly Patients With Resectable Esophageal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SichuanU
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Carboplatin; Taxes; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Carboplatin — neoadjuvant chemotherapy，2cycles.
Drug: Nab paclitaxel — neoadjuvant chemotherapy，2cycles.
Drug: Sintilimab — neoadjuvant immunotherapy，2cycles.

SUMMARY:
We intend to conduct a prospective single-arm clinical study to explore the efficacy and safety of immunochemotherapy in neoadjuvant therapy in elderly patients with advanced esophageal squamous cell carcinoma. Most previous randomized controlled studies (such as the 5010 study) have excluded older patients ≥70 years of age. However, in the real world, elderly patients with esophageal cancer account for a large number of patients, and elderly people have many complications and poor tolerance to treatment, which limits the application of synchronous chemoradiotherapy in this group. There is no standard treatment plan for patients over 70 years old, and the purpose of this study is to explore the effectiveness and safety of neoadjuvant immunochemotherapy in the treatment of this group of elderly people.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥70 years (no age limit, with super-elderly patients, such as those ≥80 years, the investigator will assess whether to include them based on the actual situation; gender is not restricted).
2. ECOG PS: 0-1 points; and G8 score ≥14 points. (Patients with G8 scores <14 points will undergo Comprehensive Geriatric Assessment (CGA), and the investigator will decide on inclusion based on the assessment results).
3. Pathologically confirmed esophageal squamous cell carcinoma.
4. No history of prior anti-tumor treatment.
5. Clinical stage is T2-4aN0M0 or T1-4aN+M0, and MDT evaluation deems the patient operable (AJCC staging eighth edition).
6. Adequate organ function:

   * Hematological tests (within 7 days, without the use of hematopoietic growth factors and transfusion): Granulocyte count ≥1.5×10^9/L, platelet count ≥80×10^9/L, hemoglobin ≥80g/L.
   * Biochemical tests: Total bilirubin ≤1.5×ULN (upper limit of normal), blood alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤2.5×ULN; creatinine clearance rate ≥60 mL/min (Cockcroft-Gault formula).
   * Coagulation function: INR or PT ≤1.5×ULN (upper limit of normal). If the subject is receiving anticoagulant therapy, PT within the designated range of anticoagulant drugs is acceptable.
   * Cardiac function assessment: Normal electrocardiogram or an abnormal electrocardiogram (deemed clinically insignificant by the investigator); cardiac Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥50%.
7. Willing to voluntarily participate in this clinical study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. Concurrent presence of other malignant tumors.
2. Active autoimmune diseases or a history of autoimmune diseases, such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (eligible after normal hormone replacement therapy).
3. Uncontrollable severe systemic diseases (involving the central nervous system, cardiovascular system, hematological system, digestive system, endocrine system, respiratory system, urogenital system, immune system, etc.) and patients with mental illness.
4. Severe cardiovascular events: heart failure (NYHA III-IV), myocardial infarction, unstable angina, severe arrhythmia, stroke, or cerebral hemorrhage within the last 6 months.
5. Congenital or acquired immunodeficiency (such as HIV infection), active hepatitis B (HBV-DNA ≥ 10^4 copies/mL) or hepatitis C (positive HCV antibodies, and HCV-RNA higher than the detection limit of the analysis method).
6. Allergy or intolerance to the investigational drug.
7. Other conditions deemed unsuitable for inclusion in this study by the investigator.

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | Within two months after surgery

SECONDARY OUTCOMES:
one-year Disease-free-survival rate | Within one year after surgery
Surgical Completion Rate | Within two months after surgery
R0 resection rate | Within two months after surgery
Incidence of Adverse events to Neoadjuvant and Surgical Treatment | From the start of treatment to three months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- West-China Hospital, Chengdu, China

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the West China Hospital of Sichuan University but restrictions apply to the availability of these data, which were used under license for the current study, and so are not publicly available. Data are however available from the authors upon reasonable request and with the permission of West China Hospital of Sichuan University. If anyone wants to request the date of the study, please contact the author, Zhen Lin. E-mail: linzhenzlk@163.com.